CLINICAL TRIAL: NCT03404492
Title: Effects of Cardiorespiratory Rehabilitation on the Right Ventricle in Pulmonary Hypertension
Acronym: Rehab-HTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-PP-09
Record Dates: First submitted 2018-01-12; First posted 2018-01-19 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with pulmonary hypertension (Other)
  Interventions: Other: Stress echocardiography

INTERVENTIONS:
Other: Stress echocardiography — A stress echocardiography will be performed in addition to the traditional patient care

SUMMARY:
Clinical improvement has been demonstrated after cardiorespiratory rehabilitation in patients with pulmonary hypertension. Rehabilitation is therefore now part of the recommendations for good practice. However, no data is available to elucidate the mechanism of this improvement: an improvement in myocardial reserve or an improvement in peripheral muscular capacity? The main objective of this study is to evaluate the difference in right ventricular contractile reserve before and after cardiorespiratory rehabilitation during stress ultrasound in pulmonary hypertension in 10 patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Major patients
* Proven pulmonary hypertension: PAPm ≥ 25mmHg, known PH
* Group 1,3,4 or 5 of the pulmonary hypertension classification
* Clinical stability > 1 month clinically determined by clinician
* NYHA II or III class
* Signature of informed consent form following appropriate information
* Patient affiliated to the Social Security System

Exclusion Criteria:

* Associated left heart disease
* Complex congenital heart disease
* Acoustic window which does not allow the echocardiography to be performed correctly
* Permanent cardiac arrhythmia
* NYHA IV class and NYHA I class
* Inability to perform at least a minimal effort on an ergometer
* Unstabilized acute coronary syndrome
* Compensatory heart failure
* Disturbances of ventricular rhythm veins, may not be narrowed.
* Prevalence of high-risk embolic intracardiac thrombus
* Prevalence of high-risk embolic intracardiac thrombus
* Preference of a medium to high abundance peericard-like thinning.
* Venous thromboembolic venous thromboembolic disease (> 3 months)
* Left ventricular ejector obstruction (severe and/or symptomatic)
* Persons under guardianship, under curatorship, protected by law
* Persons deprived of their liberty
* Pregnant and parturient women
* Major not able or unable to express consent
* Minors
* Inability to perform cardiac rehabilitation
* Modynamic instability
* Follow-up impossible for geographical or psychological reasons
* Inadequate command of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
Improvement of the subpulmonary ITS at effort >20% (presence of a right ventricular contractile reserve) defined by the improvement of the ITS or integral subpulmonary time-speed) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pamela MOCERI, PH, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hôpital Pasteur, Nice, France